CLINICAL TRIAL: NCT07367776
Title: Effects and Mechanisms of Patient Education in Osteoporosis: A Randomized Controlled Trial Comparing Digital Education, Face-to-Face Education, and General Patient Information (RCT-PATOS)
Brief Title: Patient Education in Osteoporosis (RCT-PATOS)
Acronym: RCT-PATOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Örebro County Council (Other Government); Kalmar County Council (Unknown); County Council of Halland, Sweden (Other Government); Sormland County Council, Sweden (Other); County Council of Gavleborg (Other); Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Anna Spangeus, Senior Associated Professor, Senior Consultant, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-PATOS
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis
Keywords: osteoporosis; patient education; self-care; health related quality of life; HRQoL; internetbased; digital
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Control) (Active Comparator): General information on osteoporosis (open website)
  Interventions: Behavioral: General information on osteoporosis (open website)
- Face-to-face patient education (Active Comparator): Structured group-based theoretical education ('osteoporosis school')
  Interventions: Behavioral: Face-to-face patient education
- Digital patient education (Active Comparator): Internet-based patient education program
  Interventions: Behavioral: Digital patient education

INTERVENTIONS:
Behavioral: Digital patient education — An internet-based program comprising nine modules will be available to participants for a duration of one year. The program addresses essential components of patient education in osteoporosis and includes a variety of learning formats such as text, images, videos, reflection exercises, knowledge-check questions, and checklists. The estimated total time required to complete the program is approximately 5.5 hours. Intervention adherence will be monitored. For the digital intervention, adherence will be assessed by number of modules accessed.
  Arms: Digital patient education
Behavioral: Face-to-face patient education — Three theoretical sessions, each lasting two hours, will be conducted over a period of 3-5 weeks. The sessions adhere to a standardized curriculum addressing key aspects of osteoporosis management. Two sessions will be led by physiotherapists, and one session by either a physician or a nurse. Each group will include a maximum of 15 participants. Intervention adherence will be monitored. For the group-based intervention, attendance at scheduled sessions will be recorded.
  Arms: Face-to-face patient education
Behavioral: General information on osteoporosis (open website) — Participants receive general osteoporosis information provided by healthcare services (open website with general information on osteoporosis: https://www.1177.se/sjukdomar--besvar/skelett-leder-och-muskler/benskorhet---osteoporos/ ).
  Arms: Usual care (Control)

SUMMARY:
The objective of this randomized clinical trial is to assess both the effectiveness and underlying mechanisms of patient education for individuals aged 50 years and older with osteoporosis.

Primary research question: What differences in outcomes can be observed among three different educational interventions with respect to osteoporosis-specific self-care, health related quality of life, fracture risk, illness perception, physical activity, physical function, fear of falling, and pain in patients diagnosed with osteoporosis?

The trial will include three study arms: 1) Control group: Participants receive standard osteoporosis information provided by healthcare services. 2) Face-to-face education: Three 2-hours sessions led by a physiotherapist (two sessions) and physician or nurse (one session) within a 2 months period. 3) Digital education: Internet-based program consisting of nine modules accessible to participants over a one-year period.

Participants will complete questionnaires and undergo physical assessments at baseline, and at 3 and 12 months follow up. Additionally, a subset of participants will undergo objective assessment of physical activity pattern and sedentary behaviours with an accelerometer at baseline and after 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* Age > 50 years
* Diagnosed with osteoporosis or osteopenia (either ICD-coded [M80x, M81x, or M859] or current/previous pharmacological treatment for osteoporosis)
* Basic computer literacy
* Possession of BankID (Swedish electronic identification system used for secure authentication) and ability to log in to the 1177.se "Support and Treatment platform"

Exclusion Criteria:

* Inability to understand written and spoken Swedish
* Cognitive impairment preventing comprehension of the study protocol and provision of informed consent
* Participation in structured patient education on osteoporosis within the past year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis specific self-care - OsCare Questionnaire (baseline to follow up at 12 months) | Baseline to follow up at 12 months.
  The OsCare questionnaire is a self-administered assessment designed to evaluate patients' knowledge, motivation, and behavior related to osteoporosis management. It consists of items rated on an ordinal scale, where higher values indicate more favorable responses. The instrument yields both an overall score reflecting the general level of osteoporosis-related self-care, and subscale scores corresponding to the individual domains (knowledge, motivation, and behavior).

SECONDARY OUTCOMES:
Osteoporosis specific self-care - OsCare Questionnaire (baseline to follow up at 3 months) | Baseline to follow-up at 3 months.
  The OsCare questionnaire is a self-administered assessment designed to evaluate patients' knowledge, motivation, and behavior related to osteoporosis management. It consists of items rated on an ordinal scale, where higher values indicate more favorable responses. The instrument yields both an overall score reflecting the general level of osteoporosis-related self-care, and subscale scores corresponding to the individual domains (knowledge, motivation, and behavior).
Health-related quality of life (HRQoL) - RAND-36 | Baseline to follow-up at 3 months and 12 months.
  Assessed with RAND 36-Item Health Survey. The RAND-36 compromises 36 items covering 8 health-related domains.
Health-related quality of life (HRQoL) - EQ-5D-5L | Baseline to follow-up at 3 months and 12 months.
  Assessed with the EuroQol 5 Dimensions (EQ5D-5L) and Visual Analogue Scale (VAS 0-100) where respondents rate their overall health.
Patient enablement instrument (PEI) | 3 months and 12 months
  Measured with the Patient Enablement Instrument (PEI).
Fear of falling | Baseline to follow-up at 3 months and 12 months.
  Assessed with Falls Efficacy Scale-International (FES-I). The FES-I is a 16-item questionnaire.
Illness perception | Baseline to follow-up at 3 months and 12 months.
  Assessed with the Brief-Illness Perception Questionnaire BIPQ which is an 8-item questionnaire.
Beliefs about the necessity of prescribed medication | Baseline to follow-up at 3 months and 12 months.
  Assessed using Beliefs about Medicines Questionnaire (BMQ).
Physical activity (self-reported) | Baseline to follow-up at 3 months and 12 months.
  Measured with questions from the Swedish Questionnaire about Lifestyle Habits.
Fall incidence (self-reported) | Baseline to follow-up at 3 months and 12 months.
  Self-reported numbers of fall during the last 3 and 12 months
Perceived balance (self-reported) | Baseline to follow-up at 3 months and 12 months.
  Self-rated perceived balance is assessed with Numeric Rating Scale (NRS 0-10).
Perceived pain (self-reported) | Baseline to follow-up at 3 months and 12 months.
  Self-reported pain is assessed both regarding intensity (Numeric Rating Scale [NRS] 0-10) and frequency.
Use of pain-relieving medication (self-reported) | Baseline to follow-up at 3 months and 12 months.
  Self-reported use of pain-relieving medication, including type and frequency.
Fracture risk score | Baseline to follow-up at 3 months and 12 months.
  Composite score based on results for balance (One-leg-standing test with eyes opened), leg muscle srength (Chair-Stand test- 30 sec), and patient-reported fall incidence during the last year.
Maximal walking speed | Baseline to follow-up at 3 months and 12 months.
  Walking speed assessed with patients walking 10 meters at a maximal walking speed.
Hand-strength | Baseline to follow-up at 3 months and 12 months.
  Assessed in sitting position with the Jamar. Values from both right and left side are assessed.
Chair-Stand test (30 sec) | Baseline to follow-up at 3 months and 12 months.
  The maximal number of sit to stand during 30 seconds.
Measure of hyperkyfosis | Baseline to follow-up at 3 months and 12 months.
  With patients in upright standing measuring distance between the C7 and the wall
Timed-up and go (TUG) | Baseline to follow-up at 3 months and 12 months.
  Patients were asked to stand up from sitting and walk 3 meters, turning around, walk back and sit again. Time was measured in seconds.
Static balance | Baseline to follow-up at 3 months and 12 months.
  Assessed with the One-leg-Standing test with eyes opened (OLST-EO) for both right and left legs and a maximum of 60 seconds.
Dynamic balance | Baseline to follow-up at 3 months and 12 months.
  Measured with the Four Square Step Test (FSST) as the time in seconds to perform a sequence that require the subject to step forward, backward, and sideway to the right and left.

OTHER OUTCOMES:
Accelerometer-based assessment of physical activity and sedentary behaviours | Baseline to follow-up at 3 months and 12 months.
  Measured with ActivPAL™ accelerometers in a subset of patients during 7 days
Adverse event | Baseline to follow-up at 3 months and 12 months
  Adverse events will be monitored throughout the study period. Self-reported adverse events related to fracture, musculoskeletal injury, falls, increased uncertainty and worry, or other health-related complaints will be collected at follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spångeus, Ass Prof MD, Study Chair — Region Östergötland; Johanna Wibault, PhD, Principal Investigator — Region Östergötland; Gunnel Peterson, Assoc Prof, Principal Investigator — Sormland County Council, Sweden
Locations (7):
- Sweden (7):
  - Region Gävleborg, Gävle
  - Region Jönköpings län, Jönköping
  - Region Kalmar, Kalmar
  - Region Sörmland, Katrineholm
  - Region Halland, Kungsbacka
  - Region Östergötland, Linköping
  - Region Örebro, Örebro

IPD SHARING:
Plan to Share IPD: No